CLINICAL TRIAL: NCT01861197
Title: Phase II Study of Dovitinib for FGFR1 Amplified Squamous Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Ju Ahn, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-09-070-002
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Squamous NSCLC
Keywords: Efficacy; Dovitinib; Squamous NSCLC
MeSH Terms: interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dovitinib monotherapy (Experimental)
  Interventions: Drug: Dovitinib

INTERVENTIONS:
Drug: Dovitinib — Dovitinib 500mg daily for 5 days on/ 2 day off until progression

SUMMARY:
Efficacy of Dovitinib for Squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed squamous NSCLC
* Previously treated with one or two lines of chemotherapy
* FGFR amplification (FISH > 5 copies of genes)
* 20 years or older
* ECOG PS 0-2

Exclusion Criteria:

* active infection
* uncontrolled brain metastasis
* unstable angina or MI

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
response rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Myung-Ju Ahn, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea